CLINICAL TRIAL: NCT03547258
Title: Italian Non-Interventional Study of FMS-like Tyrosine Kinase (FLT3) Mutated Acute Myeloid Leukemia (AML) Patients
Brief Title: Italian Non-Interventional Study of FLT3 Mutated AML Patients
Acronym: FLAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRST204.01
Record Dates: First submitted 2018-05-11; First posted 2018-06-06 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: AML; FLT3-ITD Mutation; FLT3-TKD Mutation
Keywords: AML; Italian observational study; FLT3-ITD Mutation; FLT3-TKD Mutation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AML patients: Clinical and Molecular data collection of AML Patients with FLT3 mutations (ITD or TKD)
  Interventions: Genetic: Clinical and Molecular data collection

INTERVENTIONS:
Genetic: Clinical and Molecular data collection — Clinical and Molecular data collection at diagnosis, during treatment and at each relapse

SUMMARY:
This is an observational study involving a retrospective and prospective collection of clinical and molecular data regarding patients with AML with FLT3+ mutations

DETAILED DESCRIPTION:
This is an observational study involving a retrospective and prospective collection of clinical and molecular data. Patients will follow their regular diagnostic and clinical practice. Thus, no additional procedure/blood withdrawal will be performed.

The study will be conducted as follows:

1. Retrospective phase: clinical and molecular data of AML patients with FLT3+ mutations detected at diagnosis or at any refractory/relapse state will be collected.
2. Prospective phase: clinical and molecular data of each new FLT3+ AML patient identified in participating centers at diagnosis or at any refractory/relapse state will be collected prospectively. Every effort will be done to include all consecutive patients, in order to avoid selection bias.

For patients with a mutation found at the time of disease relapse, any effort will be done to collect all the clinical and molecular information since the time of diagnosis.

The Primary objective of this study is to analyze how FLT3 mutational status evolve during the management of the disease looking at the percentage of patients with no FLT3 mutations at diagnosis who relapse with a new FLT3 mutation detected, and the percentage of FLT3 positive AML patients that after having obtained a Complete Remission relapse with FLT3 negative.

The secondary objective of the study is to investigate the association between different FLT3 mutations and the clinical, molecular and biological information.

ELIGIBILITY:
Inclusion criteria:

1. AML patients
2. Male or Female
3. Aged ≥ 18 years
4. FLT3 mutations (ITD or TKD) positive tests performed at diagnosis or at relapse.
5. Participant is willing and able to give informed consent for participation in the study.

Exclusion criteria:

1. To be currently involved in experimental clinical protocol, or have been treated with experimental drugs are not exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patient with FLT3 mutated AML documented at diagnosis or at the time of relapse/refractory state treated in the participating center. With regards to the retrospective collection, data from the eligible and acconsenting patients will be retrieved since 2012, that is, when the evaluation of FLT3 mutation was almost routine in the centers considered in the study.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
percentage of patients FLT3 negative at diagnosis who relapse FLT3 positive; | up to 24 months
  description of how the FLT3 mutational status changes during the course and management of the disease
percentage of patients FLT3 positive at diagnosis who relapse FLT3 negative | up to 24 months
  description of how the FLT3 mutational status changes during the course and management of the disease

SECONDARY OUTCOMES:
objective overall response rate (ORR) | up to 24 months
  the objective overall response rate (ORR) defined as the proportion of patients with a partial or response (CR, CRi, CRp) response, to initial treatment and in case of salvage;
disease-free survival (DFS) | up to 24 months
  disease-free survival (DFS) after first CR and after CR2/CR3, if applicable, defined as the time since CR (or CR2 or CR3) to disease relapse or death for any cause, whichever occurs first.
overall survival (OS) | up to 24 months
  overall survival (OS) defined as the time since date of diagnosis until death for any cause or the last available patient contact.
Percentage of AML patients with specific types of FLT3 mutations | up to 24 months
  Percentage of AML patients with specific types of FLT3 mutations, at initial diagnosis and at disease relapse
distribution of specific FLT3 mutations in AML patients | up to 24 months
  distribution of specific FLT3 mutations in AML patients according to: age, WBC, LDH, cytogenetics, NPM1, CEBPA alterations, IDH1/2, tp53, DNMT3A, secondary vs de novo AML;
frequency of the different methods used to evaluate (Minimal residual disease) MRD | up to 24 months
  the frequency of the different methods used to evaluate MRD such as, wt1 ratio or the fusion transcript level by Reverse transcription polymerase chain reaction (RT-PCR); percentage of patients performing FLT3 ITD analysis by Next Generation Sequencing (NGS);
FLT3-ITD allelic ratio | up to 24 months
  FLT3-ITD allelic ratio defined as the ratio of the area under the curve of mutant and wild type alleles (mutant/totalFLT3) obtained after Fragment analysis for FLT3-ITD;
transplantation percentage | up to 24 months
  percentage of FLT3 mutated AML patients undergoing transplantation
evaluation of modifications in terms of quality of life (QoL) of patients with FLT3 mutated AML | up to 24 months
  scores for each patient and each scale as well as a summary QoL score will be computed according to the EORTC QLQ-C3 (quality of life questionnaire) manual
retrospective collection of surrogate measures of QoL | up to 24 months
  the surrogate measures of QoL , as the number and days of hospitalizations per patient, number of clinical visits per patient, number of access in Day Hospital and Emergency Care Units per patient, and the use of antalgic drugs and neuro-active drugs, will be expressed in terms of mean values per patient or through proportions

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Martinelli, MD, Study Chair — Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST)
Locations (33):
- Italy (33):
  - AOU Ospedali riuniti di Ancona, Ancona, AN
  - AOU Policlinico Bari - Ematologia, Bari, BA
  - Università di Bologna - DIMES, Bologna, BO
  - ASST Spedali di Brescia, Brescia, BS
  - Azienda Ospedaliera G. Brotzu, Cagliari, CA
  - Azienda Ospedaliera S. Croce e Carle, Cuneo, CN
  - Ematologia - Azienda Ospedaliera "Pugliese Ciaccio" di Catanzaro, Catanzaro, CZ
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC
  - AOU Universitaria Arcispedale Sant'Anna, Cona, Ferrara
  - IRCCS Casa sollievo della sofferenza, San Giovanni Rotondo, FG
  - AOU Careggi, Florence, FI
  - Ospedale Vito Fazzi di Lecce, Lecce, LE
  - AOU Policlinico Gaetano Martino, Messina, ME
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, MI
  - Ospedale San Raffaele, Milan, MI
  - Istituto Europeo di Oncologia, Milan, MI
  - Ospedali Riuniti Villa Sofia-Cervello, Palermo, PA
  - Ospedale "Guglielmo da Saliceto", Piacenza, PC
  - Irccs Crob, Rionero in Vulture, Potenza
  - Azienda Ospedaliero-Universitaria di Parma - Ematologia e CTMO, Parma, PR
  - UO Ematologia, Ospedale S.Maria delle Croci, Ravenna, RA
  - Grande Ospedale Metropolitano, Reggio Calabria, RC
  - Ospedale infermi di Rimini, Rimini, RN
  - AOU San Giovannidi Dio e Ruggi - ematologia, Salerno, SA
  - AOC di Ematologia - AOU Senese, Siena, SI
  - Università di Torino - Ospedale San Luigi Gonzaga, Orbassano, TO
  - AOU Città della Salute e della Scienza di Torino, Torino, TO
  - A.O. Ordine Mauriziano Torino, Torino, TO
  - Divisione di Ematologia - Università di Udine, Udine, UD
  - AO Universitaria Federico II, Napoli
  - AOU Maggiore della carità, Novara
  - AOU Santa Maria della Misericordia - Ematologia, Perugia
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma